CLINICAL TRIAL: NCT00403429
Title: Phase II Study With Capecitabine as Monotherapy in the Treatment of Platinum Resistant or Refractory Ovarian Cancer.
Brief Title: MITO-6: Capecitabine in Platinum Resistant Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MITO-6; EudraCT number 2006-001724-40
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Ovarian Cancer
Keywords: oral chemotherapy; platinum resistant; platinum refractory; second line
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Capecitabine

ARMS (1):
- Capecitabine (Experimental)
  Interventions: Drug: capecitabine

INTERVENTIONS:
Drug: capecitabine

SUMMARY:
The purpose of this study is to evaluate the activity and the toxicity of capecitabine as monotherapy in the treatment of platinum resistant or refractory ovarian cancer.

DETAILED DESCRIPTION:
Ovarian cancer is the second most frequent and the most deadly gynaecologic cancer. Standard combination chemotherapy with a platinum derivative (cisplatin or carboplatin) and a taxane are effective in causing remission in 60 - 80 % of cases, yet recurrences are frequent and 5-year survival is only 20%. Current therapies for second line treatment of recurrence in patients who have platinum refractory (who experienced progression of the disease during first line platinum based therapy) or platinum resistant (who experienced a recurrence of the disease within 6 months of completing platinum based therapy)ovarian cancer are limited. Capecitabine, an oral chemotherapy already used in colon and breast cancers, has shown some promise in early clinical trials for treating recurrent ovarian cancer.

Patients entered into this trial will receive oral capecitabine 1250 mg/m2 on days 1-14 every 21 days for up to 6 cycles, depending on response.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histologic diagnosis of relapsed ovarian cancer
* Refractory or resistant to platinum salts disease
* Age < 75 years
* At least one measurable lesion (³ 20 mm with conventional techniques or ³ 10 mm with spiral CT scan)
* Life expectancy of at least 3 months
* Written informed consent

Exclusion Criteria:

* Previous or concomitant malignant neoplasia within 5 years prior to basal evaluation (excluding adequately treated basocellular or spinocellular skin carcinoma or in situ carcinoma of the uterine cervix).
* Performance Status (ECOG) ³ 3
* Previous chemotherapy treatment with capecitabine
* More than 3 lines of chemotherapy
* Heart disease (heart failure, heart attack during the 6 months prior to the trial, atrioventricular block of any degree, serious arrhythmia)
* Leukocytes < 4000/mm3, platelets < 100000/mm3
* Modifications of renal function (Creatinine ³ 1.25 times the upper normal limit) or liver function (SGOT or SGPT ³ 1.25 times the upper normal limit)
* Present or suspected haemorrhagic syndromes
* Uncooperative and/or unreliable patients
* Patients' inability to access the centre

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-03; Primary Completion 2008-01 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
objective response rate | 6 months
toxicity | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Ph.D, Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute, Naples
Locations (17):
- Italy (17):
  - Clinica Malzoni, Reparto di Ginecologia Oncologica, Avellino, AV
  - Ospedale Regionale Miulli, Divisione Medicina Interna Sezione Oncologica, Acquaviva delle Fonti, BA
  - IRCCS Oncologico Bari, Oncologia Medica, Bari, BA
  - Ospedale Fatebenefratelli, U.O. di Oncologia, Benevento, BN
  - Ospedale Cannizzaro, Divisione di Ostetricia e Ginecologia, Catania, CT
  - IRCCS Casa Solllievo della Sofferenza, San Giovanni Rotondo, FG
  - Azienda Ospedaliera Carlo Poma, Divisione di Oncologia ed Ematologia, Mantova, MN
  - Ospedale Ramazzini, Day Hospital Oncologico, Carpi, MO
  - Policlinico Universitario P. Giaccone, Palermo, PA
  - Casa di Cura La Maddalena S.p.A., Dipartimento Oncologico, Palermo, PA
  - Ospedale S. Massimo, Day Hospital Oncologico, Penne, PE
  - Centro di Riferimento Oncologico, Divisione di Oncolgia Medica C, Aviano, PN
  - Azienda Ospedaliera S. Maria degli Angeli, Servizio di Oncologia, Pordenone, PN
  - Ospedale S. Giovanni Calibita Fatebenefratelli, Roma, Roma
  - Ospedale S. Bortolo ULSS 6, U.O. di Oncologia Medica, Vicenza, VI
  - Istituto Nazionale dei Tumori , Divisione di Oncologia Medica B, Napoli
  - Istituto Nazionale dei Tumori, Divisione di Oncologia Medica C, Napoli

REFERENCES:
- [Result] Pisano C, Morabito A, Sorio R, Breda E, Lauria R, Gebbia V, Scaltriti L, Scalone S, Zagonel V, Greggi S, Beneduce G, Losito S, Gallo C, Di Maio M, Forestieri V, Pignata S. A phase II study of capecitabine in the treatment of ovarian cancer resistant or refractory to platinum therapy: a multicentre Italian trial in ovarian cancer (MITO-6) trial. Cancer Chemother Pharmacol. 2009 Oct;64(5):1021-7. doi: 10.1007/s00280-009-0958-0. Epub 2009 Mar 6. PMID 19266200